CLINICAL TRIAL: NCT03016351
Title: Improving Blood Pressure and Cardiovascular Risk With Resistance Exercise in African Americans
Acronym: BPVR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Shane Phillips, PT, PhD, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1091; R01HL130513-01A1 (NIH)
Record Dates: First submitted 2017-01-06; First posted 2017-01-10 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Hypertension; Cardiovascular Diseases; Vascular Diseases
Keywords: Hypertension; Exercise; African Americans; Arterial Function; Arterial Stiffness
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Vascular Diseases; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aerobic Training (Experimental): Participants will undergo a supervised endurance training program in accordance with established guidelines. Each session will be monitored by a physical therapist or exercise physiologist. Sessions will be carried out 3 times per week. During each session, participants will complete a 5 min warm-up followed by 30-45 min of endurance exercise using cycle ergometry. Intensity will be monitored using heart rate monitors during each exercise session, and each participant will receive an exercise prescription with a heart range equivalent to 65-85% of their heart rate max. Participants will be asked to complete 30 min of exercise during each session in week 1, 35 min in week 2 and 40-45 min weeks 3-8 with a 5 min cool down period.
  Interventions: Other: Aerobic Training
- Resistance Training (Experimental): Participants will undergo a supervised resistance training program in accordance with established guidelines. Each session will be monitored by a physical therapist or exercise physiologist. Sessions will be carried out 3 times per week, 45 min per session. Muscle strength will be determined once before and once after resistance training by measuring ten repetition maximum (10 RM) for each exercise. Eight exercises (three sets; 8-12 repetitions) will be used on each of the large muscle groups (leg press, leg extension, leg curl, chest press, shoulder extension, biceps curl, abdominal crunch and back extension). In addition, workloads will be progressively increased if the patients can lift the weight more than 12 repetitions.
  Interventions: Other: Resistance Training

INTERVENTIONS:
Other: Aerobic Training — After the subject meets all inclusion and exclusion criteria, the subject will be randomized equally to either the ResistanceTraining group (RT) or Aerobic Training group (AT) for weeks 9-16 of the intervention. The participants will be supervised by physical therapists and/or exercise physiologists. Sessions will occur 3 days a week and will be 45 minutes in duration.
  Arms: Aerobic Training
Other: Resistance Training — After the subject meets all inclusion and exclusion criteria, the subject will be randomized equally to either the ResistanceTraining group (RT) or Aerobic Training group (AT) for weeks 9-16 of the intervention. The participants will be supervised by physical therapists and/or exercise physiologists. Sessions will occur 3 days a week and will be 45 minutes in duration.
  Arms: Resistance Training

SUMMARY:
After the participant meets all inclusion and exclusion criteria, they will be randomized equally to either the Resistance Training group (RT) or Aerobic Training group (AT). Both groups will participate in an 8 week initial control period, followed by 8 weeks of supervised exercise training, followed by 8 weeks of deconditioning. All participants will undergo the same assessments and procedures one time prior to the initial 8 week control period, and at each of the three periods. Assessments include: blood draws; arterial stiffness testing; ultrasounds of the brachial artery to measure flow-mediated dilation (FMD); gluteal adipose tissue biopsies; exercise testing to determine VO2 max; body composition analysis via DEXA scans; ambulatory blood pressure measurement; diet analysis via food journals; medical history questionnaires; urine analysis for pregnancy; and activity monitoring via accelerometer. Total participation will be 24-26 weeks.

DETAILED DESCRIPTION:
This study is divided into three separate 8-week periods, the Control period, the Exercise Training period and the De-training period. Testing sessions will be done at Week 0, Week 8, Week 16, and Week 24 of the study.

Control Period (weeks 0-8): Participants will have a control period of 8 weeks. Participants will be given a brochure regarding the benefits of regular exercise and nutrition on overall health.

1. Baseline visit and eligibility assessment, Week 0: After an initial phone interview to screen participants for eligibility, participants will be scheduled for their two sessions of baseline assessments.

   Randomization After the subject meets all inclusion and exclusion criteria, the participant will be randomized equally to either the Resistance Training group (RT) or Aerobic Training group (AT) with a table of random numbers by a staff member having no knowledge of the participant's baseline profile.

   V1A (2 hours): Clinical Research Center and/or Integrative Physiology Lab

   Participants will report to the UIC CRC or UIC Integrative Physiology Lab after a 12 hour fast. Everyone will be instructed to take all prescribed medications as normal and to continue to drink plenty of water. Participants will also be told not to exercise for 24 hours prior to the testing session. Female participants will be in the follicular stage of their menstrual cycle. After informed consent and a medical history obtained, the following procedures will be performed:
   * Urine pregnancy test for women
   * Questionnaires (Health History Questionnaire, Pittsburgh Sleep Quality Index (PSQI), Physical Activity Questionnaire, Automated Self-Administered 24-hour Dietary Assessment Tool (ASA 24), and Alcohol Intake Questionnaire (AIQ)
   * Anthropometrics: weight, height, waist circumference and BMI
   * Vitals: Blood pressure and heart rate
   * Blood draw of approximately 2 tablespoons or 30 mLs
   * Arterial stiffness test via pulse wave velocity: Sphygmocor (SphygmoCor, AtCor Medical, Sydney, Australia) is a device that used to detect the stiffness of blood vessels.
   * Ultrasound for brachial flow-mediated dilation with administration of nitroglycerin
   * Beginning of 24 hour blood pressure monitoring.

   V1B (2 hours): Integrative Physiology Lab

   Participants will report to the IPL for the following procedures:
   * Exercise testing: Maximal oxygen consumption will be evaluated using the treadmill to exhaustion.
   * Dual Energy X-ray Absorptiometry (DEXA)
   * Begin 7 days of activity monitoring with accelerometer. V1C (5 minutes): Integrative Physiology Lab

   Participants will report to the IPL for the following procedures:

   • Return the accelerometer after 7 days of activity monitoring.

   Exercise Training Period (weeks 9-16): Participants will participate 3 days a week in either the Resistance Training group (RT) or the Aerobic Training group (AT).
2. Pre-training Testing, Week 8: After the 8 week control period, before training begins, participants will report for two testing visits, and will undergo the following procedures:

   V2A (2 hours): Clinical Research Center and/or Integrative Physiology Lab: Same as V1A procedures as outlined in the Baseline visit (including the 12 hour fast), with the addition of a subcutaneous gluteal fat biopsy that will be performed in conjunction with the above measures, or scheduled separately at the Clinical Research Center.

   V2B (2 hours): Integrative Physiology Lab: Participants will report to the IPL for the same procedures as outlined in the Baseline visit (V1B).

   V2C (5 minutes): Integrative Physiology Lab: Participants will report to the IPL for the same procedures as outlined in the Baseline visit (V1C).

   Exercise Intervention Groups:

   Aerobic Training Intervention (weeks 9-16): Subjects will undergo a supervised endurance training program in accordance with established guidelines.

   Resistance Training Intervention (weeks 9-16): Subjects randomized to 8-week resistance exercise training program will visit the UIC Integrative Physiology exercise research laboratory 3 times per week, 45 min per session.
3. Post training Testing, Week 16: The two visit post-training testing will start 24-48 hours after last exercise session to avoid potential effects of the acute exercise bout. This testing is identical to the testing that occurred at the beginning of the exercise training period (V2) at Week 8. Participants will report for two testing visits, and will undergo the following procedures:

   V3A (2 hours): Clinical Research Center and/or Integrative Physiology Lab: Same V2A procedures as outlined in the Pre-Training visit (V2A) (including the 12 hour fast).

   V3B (2 hours): Integrative Physiology Lab: Participants will report to the IPL for the same procedures as outlined in the Pre-Training visit (V2B).

   V3C (5 minutes): Integrative Physiology Lab Participants will report to the IPL for the same procedures as outlined in the Pre-Training visit (V2C).

   De-Training Follow-up (weeks 16- 24):

   All subjects will be asked to resume normal activities after the 8-week exercise training program.
4. Post-Detraining Testing, Week 24: All of the procedures described in Post-Training visits will be repeated. Participants will report for two testing visits, and will undergo the following procedures:

V4A (2 hours): Clinical Research Center and/or Integrative Physiology Lab: Same V2A procedures as outlined in the Pre-Training visit (V2A) (including the 12 hour fast).

V4B (2 hours): Integrative Physiology Lab: Participants will report to the IPL for the same procedures as outlined in the Pre-Training visit (V2B).

V4C (5 minutes): Integrative Physiology Lab Participants will report to the IPL for the same procedures as outlined in the Pre-Training visit (V2C).

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* Body Mass Index of 18.5-40 kg/m²
* Born in the United States of either two African-American or two non-Hispanic Caucasian parents
* Blood pressure of at least 120/80 mmHg

Exclusion Criteria:

* Inability to give informed consent
* History of cardiovascular disease or cardiovascular events
* Hypertension (systolic >159 mmHg and diastolic >99 mmHg) or on more than one anti-hypertensive medication
* Diabetes Type I& II
* Hyperlipidemia, with an LDL-C >159 mg/dL and /or total-C >229 mg/dL
* Pregnancy (or intend to become pregnant while participating in study) or nursing
* Tobacco use in the past 6 months (including, but not limited to cigarettes, e-cigarettes, hookah, Nicorette, SNUs and chewing tobacco)
* Chronic inflammatory disease such as, but not limited to, cancer
* Chronic autoimmune diseases such as, but not limited to: lupus, multiple sclerosis, rheumatoid arthritis
* Adverse reaction to nitroglycerin
* Anemia with a hemoglobin < 8
* Head injury within last 6 months
* Seizure disorder
* Presence of renal disease with a creatinine > 1.5mg/dL
* Presence of liver disease with liver enzymes > 3x the upper limits of normal
* Currently abusing alcohol or illicit drugs
* Unreliability as a study subject, in the opinion of the Investigator
* Lidocaine allergy
* Amenorrhea
* Postmenopausal women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2016-10; Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Changes in peripheral and central blood pressure | Baseline (wk. 0), Pre-training (wk. 8), post- training (wk. 16), post detraining (wk. 24)

SECONDARY OUTCOMES:
Changes in arterial stiffness | Baseline (wk. 0), Pre-training (wk. 8), post- training (wk. 16), post detraining (wk. 24)
Changes in endothelial function | Baseline (wk. 0), Pre-training (wk. 8), post- training (wk. 16), post detraining (wk. 24)

CONTACTS AND LOCATIONS:
Overall Officials: Shane Phillips, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):143-52. doi: 10.1161/CIR.0b013e318282ab8f. No abstract available. PMID 23283859
- [Result] Ogedegbe G, Tobin JN, Fernandez S, Cassells A, Diaz-Gloster M, Khalida C, Pickering T, Schwartz JE. Counseling African Americans to Control Hypertension: cluster-randomized clinical trial main effects. Circulation. 2014 May 20;129(20):2044-51. doi: 10.1161/CIRCULATIONAHA.113.006650. Epub 2014 Mar 21. PMID 24657991
- [Result] Fields LE, Burt VL, Cutler JA, Hughes J, Roccella EJ, Sorlie P. The burden of adult hypertension in the United States 1999 to 2000: a rising tide. Hypertension. 2004 Oct;44(4):398-404. doi: 10.1161/01.HYP.0000142248.54761.56. Epub 2004 Aug 23. PMID 15326093
- [Result] Zion AS, Bond V, Adams RG, Williams D, Fullilove RE, Sloan RP, Bartels MN, Downey JA, De Meersman RE. Low arterial compliance in young African-American males. Am J Physiol Heart Circ Physiol. 2003 Aug;285(2):H457-62. doi: 10.1152/ajpheart.00497.2002. Epub 2003 May 8. PMID 12738618
- [Result] Kaess BM, Rong J, Larson MG, Hamburg NM, Vita JA, Levy D, Benjamin EJ, Vasan RS, Mitchell GF. Aortic stiffness, blood pressure progression, and incident hypertension. JAMA. 2012 Sep 5;308(9):875-81. doi: 10.1001/2012.jama.10503. PMID 22948697
- [Result] Heffernan KS, Jae SY, Wilund KR, Woods JA, Fernhall B. Racial differences in central blood pressure and vascular function in young men. Am J Physiol Heart Circ Physiol. 2008 Dec;295(6):H2380-7. doi: 10.1152/ajpheart.00902.2008. Epub 2008 Oct 10. PMID 18849329
- [Result] Vita JA. Nitric oxide and vascular reactivity in African American patients with hypertension. J Card Fail. 2003 Oct;9(5 Suppl Nitric Oxide):S199-204; discussion S205-9. doi: 10.1054/s1071-9164(03)00588-8. No abstract available. PMID 14583889
- [Result] Heffernan KS, Fahs CA, Iwamoto GA, Jae SY, Wilund KR, Woods JA, Fernhall B. Resistance exercise training reduces central blood pressure and improves microvascular function in African American and white men. Atherosclerosis. 2009 Nov;207(1):220-6. doi: 10.1016/j.atherosclerosis.2009.03.043. Epub 2009 Apr 5. PMID 19410255
- [Result] Franzoni F, Ghiadoni L, Galetta F, Plantinga Y, Lubrano V, Huang Y, Salvetti G, Regoli F, Taddei S, Santoro G, Salvetti A. Physical activity, plasma antioxidant capacity, and endothelium-dependent vasodilation in young and older men. Am J Hypertens. 2005 Apr;18(4 Pt 1):510-6. doi: 10.1016/j.amjhyper.2004.11.006. PMID 15831361
- [Result] Sato A, Miura H, Liu Y, Somberg LB, Otterson MF, Demeure MJ, Schulte WJ, Eberhardt LM, Loberiza FR, Sakuma I, Gutterman DD. Effect of gender on endothelium-dependent dilation to bradykinin in human adipose microvessels. Am J Physiol Heart Circ Physiol. 2002 Sep;283(3):H845-52. doi: 10.1152/ajpheart.00160.2002. PMID 12181110
- [Result] Williams MR, Westerman RA, Kingwell BA, Paige J, Blombery PA, Sudhir K, Komesaroff PA. Variations in endothelial function and arterial compliance during the menstrual cycle. J Clin Endocrinol Metab. 2001 Nov;86(11):5389-95. doi: 10.1210/jcem.86.11.8013. PMID 11701712
- [Result] Hashimoto M, Akishita M, Eto M, Ishikawa M, Kozaki K, Toba K, Sagara Y, Taketani Y, Orimo H, Ouchi Y. Modulation of endothelium-dependent flow-mediated dilatation of the brachial artery by sex and menstrual cycle. Circulation. 1995 Dec 15;92(12):3431-5. doi: 10.1161/01.cir.92.12.3431. PMID 8521564
- [Result] Ling C, Diaz KM, Kretzschmar J, Feairheller DL, Sturgeon KM, Perkins A, Veerabhadrappa P, Williamson ST, Lee H, Grimm H, Babbitt DM, Brown MD. Chronic aerobic exercise improves blood pressure dipping status in African American nondippers. Blood Press Monit. 2014 Dec;19(6):353-8. doi: 10.1097/MBP.0000000000000075. PMID 25100263